CLINICAL TRIAL: NCT03513419
Title: The AMOR Method: Resilience Training for Parents of Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45774
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMOR Method (Experimental): The AMOR Method: The parent resilience training involves a series of eight weekly 90-minute group sessions, as well as three individual sessions. Group session content includes training in mindfulness, grief and loss processing, acceptance and committed actions, optimistic thinking, and resilience through the use of didactic training, group discussions, and homework assignments. Individual session content will center on additional and individualized training in grief and loss processing, optimistic thinking, and maintaining resilience over time.
  Interventions: Behavioral: The AMOR Method
- Wait List (No Intervention): Participants assigned to the waitlist will continue stable treatments and will be offered the opportunity to participate in the treatment after completion of the 8-week trial.

INTERVENTIONS:
Behavioral: The AMOR Method — The parent resilience training involves a series of eight weekly 90-minute group sessions with up to 8 parents of young children with ASD (4- 10:11 years old) per group, as well as three individual sessions.
  Arms: AMOR Method

SUMMARY:
We will evaluate whether a resilience training program which includes group and individual parent training will be effective in improving optimism and resiliency in parents of young children with autism spectrum disorders (ASD). By observing the level of parent optimism and resiliency before and after intervention, we will be able to determine whether the intervention is effective in improving parent resilience.

ELIGIBILITY:
Inclusion Criteria:

Parents eligible to participate include parents: a) English-speaking, b) of a child aged 4:0 to 10:11 years, c) with a previous diagnosis of ASD and evidence of current social impairment (SRS-2) and repetitive behaviors (RBS-R), and d) who are able to consistently participate in sessions. Given budgetary constraints, direct diagnostic testing will not be feasible. Instead, child diagnostic status will be confirmed through review of the child's medical record for evidence that the child previously met ADOS criteria for ASD and shows clinically significant social impairment at baseline (SRS-2 T>65).

Parents who are not eligible to participate include parents: a) with severe psychiatric, genetic, or medical disorder among parents and/or children, b) taking psychiatric medication, and c) with elevated resilience scores at baseline (Total Score >80 on CD-RISC). The DSM-5 CCSM will be administered to parents to screen for parent mental illness. Any identified issues on the DSM-5 CCSM will be investigated further by the PI to rule out severe psychiatric disorders.

Exclusion Criteria:

a) Severe psychiatric, genetic, or medical disorder among parents and/or children, b) parents taking psychiatric medication, and c) parents with elevated resilience scores at baseline (Total Score>80 on CD-RISC). The DSM-5 Cross Cutting Symptom Measure (DSM-5 CCSM) will be administered to parents to screen for parent mental illness. Any identified issues on the DSM-5 CCSM will be investigated further by the PI to rule out severe psychiatric disorders. These families will be referred for behavioral consultation (available in our clinic) and then be reconsidered for group participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Connor-Davidson Resilience Scale (CDRISC) from Baseline to week 8 | Baseline, week 8
  No subscales, total score only, 25 items total, 0-4 Likert Score Range: 0-100 Low resilience score (PTSD & grief populations) = 45 or lower; Average/Normal resilience score (general population) = 45-80; High Average/Elevated resilience score (yogi & meditation teachers) = 81-100 Higher total scores reflect higher levels of resilience.

SECONDARY OUTCOMES:
Change in Acceptance and Action Questionnaire-II (AAQ-II) from Baseline to week 8 | Baseline, week 8
  No subscales, total score only, 10 items total (3 items reverse scored) Score Range: 0-70 Low acceptance 0-22, Medium 23-47, High 48-70 Higher total scores reflect higher levels of optimism.
Change in Mindful Attention Awareness Scale (MAAS) from Baseline to week 8 | Baseline, week 8
  No subscales, total score only, 15 items total Score Range: 15-90 Low mindfulness score = 30 or lower; Average/Normal mindfulness score = 30-45-60; High Average/Elevated mindfulness score = 60 or higher Higher total scores reflect higher levels of dispositional mindfulness.
Change in Life Orientation Test Revised (LOT-R) from Baseline to week 8 | Baseline, week 8
  No subscales, total score only, 10 items total Score Range: 0-24 Low optimism 0-8, Medium/Average Optimism 9-16, High Optimism 17-24 Higher total scores reflect higher levels of optimism.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartzman JM, Millan ME, Uljarevic M, Gengoux GW. Resilience Intervention for Parents of Children with Autism: Findings from a Randomized Controlled Trial of the AMOR Method. J Autism Dev Disord. 2022 Feb;52(2):738-757. doi: 10.1007/s10803-021-04977-y. Epub 2021 Mar 28. PMID 33774741